CLINICAL TRIAL: NCT06555237
Title: MEK Inhibitors for the Treatment of Hypertrophic Cardiomyopathy in Patients With RASopathies (MEKinRAS) - Randomized Controlled Trial
Brief Title: MEK Inhibitors for the Treatment of Hypertrophic Cardiomyopathy in Patients With RASopathies
Acronym: MEKinRAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB/16/2024
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cardiomegaly; Noonan Syndrome
Keywords: Noonan syndrome; MEK kinase; RASOpathies; Children; Cardiomyopathy
MeSH Terms: conditions — Cardiomegaly; Noonan Syndrome; Cardiomyopathies | interventions — trametinib; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trametynib (Experimental): Trametynib in 0,025mg/kg dose orally once daily
  Interventions: Drug: Trametinib tablet
- Standard therapy (Active Comparator): Disopiramide and Beta-blocker orally
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Trametinib tablet — Trametynib orally once daily in 0,025mg/kg dose
  Arms: Trametynib
Drug: Standard therapy — Disopiramide and Beta blockers orally
  Arms: Standard therapy

SUMMARY:
The goal of this study is to evaluate the effectiveness of trametinib treatment in patients with Hyperthropic cardiomyopathy and a genetic mutation in the RAS/MAPK pathway.

DETAILED DESCRIPTION:
Introduction RASopathies are a group of genetic diseases caused by mutations in the mitogen-activated kinase (RAS-MAPK) pathway. These mutations affect many processes and are the cause of numerous genetic syndromes (including Noonan syndrome) in the course of which severe hypertrophic cardiomyopathy (HCM) develops. MEK kinase inhibitors are used to treat cancers with mutations in the RAS-MAPK pathway in adults. So far, single cases of HCM treatment in patients with RASopathies have been described, with rapid improvement in both laboratory and echocardiographic parameters and regression of myocardial hypertrophy. Due to the described effectiveness, it is reasonable to verify these effects in a well-designed randomized study on a large group of patients.

Objective To evaluate the effectiveness of trametinib treatment in patients with HCM and a genetic mutation in the RAS/MAPK pathway.

Methodology

Randomized, open-label study. The study will include patients aged 0 to 18 with:

* mutation in the RAS/MAPK pathway confirmed by genetic tests
* HCM diagnosed by echocardiography

In the first phase of the study (3 months), patients will be randomly assigned to one of two groups:

* the intervention group will receive trametinib and standard treatment (beta-blocker and disopyramide)
* the control group will receive only standard treatment. Once this phase is complete, patients will be assessed. If higher effectiveness is demonstrated in the intervention group, in the second phase of the study, patients in the intervention group will continue their current treatment and patients in the control group will receive trametinib treatment. Each group will receive trametinib for 12 months.

Importance of the study The study results will provide grounds for routine introduction of MEK kinase inhibitors for the treatment of patients with HCM due to RASopathy. If effectiveness is demonstrated, this group will gain a simple, non-invasive and causal treatment option.

ELIGIBILITY:
Inclusion Criteria:

* patient with diagnosed RASopathy
* patient with diagnosed hypertrophic cardiomyopathy
* signed innform consent

Exclusion Criteria:

* contraindications to treatment with propranolol (drug hypersensitivity, atrioventricular block, severe bradycardia) disopyramide (drug hypersensitivity, WPW syndrome, atrioventricular block, QT prolongation) trametinib (drug hypersensitivity)
* lack of consent of the child's guardians to participate in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the trametynib treatment on cardiac hyperthropy | 1 year
  Reduction of cardiac hypertrophy and/or LVOTO at 6 and 12 months of treatment and at 3 months of follow-up after treatment discontinuation using echocardiographic examination.
Effectiveness of the trametynib treatment on laboratory enzymes levels | 1 year
  Decrease in cardiac enzyme levels (NT-pro-BNP and high-sensitivity troponin I) determined in the 6th and 12th month of treatment and in the 3rd month of observation after its discontinuation.

SECONDARY OUTCOMES:
MEK kinase activity | 6 months
  Assessment of MEK kinase activity before treatment and after 6 months of its duration, in the patients' blood samples
Effectivness of the trametynib treatment assessed in the cardia magnetic resonance | 1 year
  reduction of cardiac hypertrophy in magnetic resonance imaging in the age group of 7-18 years not requiring general anesthesia (comparison of results before inclusion in the study, after 12 months of trametinib treatment and after the end of follow-up after its discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: MAciej Kołodziej, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Brouchoven I, Lorand J, Bofferding L, Sorlin A, Van Damme A, Danhaive O. Trametinib as a targeted treatment in cardiac and lymphatic presentations of Noonan syndrome. Front Pediatr. 2025 Feb 18;13:1475143. doi: 10.3389/fped.2025.1475143. eCollection 2025. PMID 40041314